CLINICAL TRIAL: NCT00678379
Title: Pediatric Tonsillectomy Pain Reduction Study, a Randomized, Placebo Controlled, Double-Blind Clinical Trial Using Clonidine and Local Anesthetics
Brief Title: Pediatric Tonsillectomy Pain Reduction Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan R. Moss, Resident Physician, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 080127
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Pain
Keywords: Tonsillectomy; Postoperative Pain; Clonidine; Anesthetics, Local
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Bupivacaine; Saline Solution; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal Saline (Placebo Comparator): 1.5 ml injection of Normal Saline into each tonsillar fossa pre-tonsillectomy
  Interventions: Drug: Normal saline
- Lidocaine (1%) + Bupivacaine 0.5% (Active Comparator): Submucosal injection of 1.5 mL Lidocaine (1%) + Bupivacaine 0.5% into the tonsillar fossa, pre-tonsillectomy
  Interventions: Drug: lidocaine (1%) + bupivacaine (0.5%)
- Lidocaine + Bupivacaine + Clondine (Experimental): Submucosal injection of 1.5 mL Lidocaine 1% + Bupivacaine 0.5% + Clondine 25mcg into the tonsillar fossa, pre-tonsillectomy
  Interventions: Drug: Lidocaine (1%) + Bupivacaine (0.5%) + Clonidine (25mcg)

INTERVENTIONS:
Drug: lidocaine (1%) + bupivacaine (0.5%) — Submucosal injection of 1.5 mL into each tonsillar fossa prior to performing tonsillectomy.
  B - lidocaine (1%) + bupivacaine (0.5%)
  Arms: Lidocaine (1%) + Bupivacaine 0.5%
Drug: Normal saline — Submucosal injection of 1.5 mL into each tonsillar fossa prior to performing tonsillectomy.
  A - normal saline
  Arms: Normal Saline
Drug: Lidocaine (1%) + Bupivacaine (0.5%) + Clonidine (25mcg) — Submucosal injection of 1.5 mL into each tonsillar fossa prior to performing tonsillectomy.
  C - lidocaine (1%) + bupivacaine (0.5%) + clonidine (25mcg)
  Arms: Lidocaine + Bupivacaine + Clondine

SUMMARY:
Tonsillectomy is associated with a significant decrease quality of life in children secondary to pain, which is worsened with swallowing. The objective of the current study is to conduct a prospective, double-blind, placebo-controlled, randomized clinical trial using a pre-tonsillectomy infiltration of the tonsillar fossa comparing three treatment regimens in reducing post-tonsillectomy morbidity (i.e. pain, poor oral intake): 1) Placebo (saline injection) 2) bupivacaine (0.5%) + lidocaine (1%), 3) bupivacaine (0.5%) + lidocaine (1%) + clonidine (25 µg).

DETAILED DESCRIPTION:
Tonsillectomy is associated with a significant decrease quality of life in children secondary to pain, which is worsened with swallowing. Previous studies in the pediatric population have demonstrated a significant decrease in post-operative pain/morbidity when administering pain reduction medications into the tonsillar fossa prior to removal. While these studies have shown great promise, no large randomized trial of the most promising medications has been conducted. Because of this, many otolaryngologists do not administer intra-operative medications aimed at reducing post-operative pain. The objective of the current study is to conduct a prospective, double-blind, placebo-controlled, randomized clinical trial using a pre-tonsillectomy infiltration of the tonsillar fossa comparing three treatment regimens in reducing post-tonsillectomy morbidity (i.e. pain, poor oral intake): 1) Placebo (saline injection) 2) bupivacaine (0.5%) + lidocaine (1%), 3) bupivacaine (0.5%) + lidocaine (1%) + clonidine (25 µg).

ELIGIBILITY:
Inclusion Criteria:

* Age 3 - 17 years old
* BMI < 35
* Negative pregnancy test in female patients age 10 and older
* Diagnosed with adenotonsillar hypertrophy, recurrent adenotonsillitis or upper airway obstruction and will be undergoing tonsillectomy alone or adenotonsillectomy

Exclusion Criteria:

* Diagnosis of obstructive sleep apnea
* Patient with peritonsillar abscess
* Allergy to study medication
* Any major systemic illness, genetic disorder or diagnosed syndrome
* Bleeding disorder

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Moss, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Monroe Carrel Jr. Children's Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share unless specifically requested within 5 year storage of data period.

REFERENCES:
- [Background] Cucchiaro G, Ganesh A. The effects of clonidine on postoperative analgesia after peripheral nerve blockade in children. Anesth Analg. 2007 Mar;104(3):532-7. doi: 10.1213/01.ane.0000253548.97479.b8. PMID 17312203
- [Background] Naja MZ, El-Rajab M, Kabalan W, Ziade MF, Al-Tannir MA. Pre-incisional infiltration for pediatric tonsillectomy: a randomized double-blind clinical trial. Int J Pediatr Otorhinolaryngol. 2005 Oct;69(10):1333-41. doi: 10.1016/j.ijporl.2005.03.020. Epub 2005 Apr 22. PMID 16159655
- [Background] McCartney CJ, Duggan E, Apatu E. Should we add clonidine to local anesthetic for peripheral nerve blockade? A qualitative systematic review of the literature. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):330-8. doi: 10.1016/j.rapm.2007.02.010. PMID 17720118
- [Background] Jebeles JA, Reilly JS, Gutierrez JF, Bradley EL Jr, Kissin I. Tonsillectomy and adenoidectomy pain reduction by local bupivacaine infiltration in children. Int J Pediatr Otorhinolaryngol. 1993 Jan;25(1-3):149-54. doi: 10.1016/0165-5876(93)90048-8. PMID 8436459
- [Background] Jebeles JA, Reilly JS, Gutierrez JF, Bradley EL Jr, Kissin I. The effect of pre-incisional infiltration of tonsils with bupivacaine on the pain following tonsillectomy under general anesthesia. Pain. 1991 Dec;47(3):305-308. doi: 10.1016/0304-3959(91)90220-R. PMID 1784501
- [Background] Giannoni C, White S, Enneking FK, Morey T. Ropivacaine with or without clonidine improves pediatric tonsillectomy pain. Arch Otolaryngol Head Neck Surg. 2001 Oct;127(10):1265-70. doi: 10.1001/archotol.127.10.1265. PMID 11587610
- [Derived] Moss JR, Cofer S, Hersey S, Goudy S, Werkhaven J, Swanson E, Mantle C, Stowell N, Byrne D, Wang L, Labadie R. Comparison of clonidine, local anesthetics, and placebo for pain reduction in pediatric tonsillectomy. Arch Otolaryngol Head Neck Surg. 2011 Jun;137(6):591-7. doi: 10.1001/archoto.2011.45. Epub 2011 Mar 21. PMID 21422302

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline: Normal Saline
  normal saline: Submucosal injection of 1.5 mL into each tonsillar fossa prior to performing tonsillectomy with one of three injections.
  A - normal saline
- Lidocaine (1%) + Bupivacaine 0.5%: Lidocaine (1%) + Bupivacaine 0.5%
  lidocaine + bupivacaine: Submucosal injection of 1.5 mL into each tonsillar fossa prior to performing tonsillectomy with one of three injections.
  B - lidocaine (1%) + bupivacaine (0.5%)
- Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg: Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
  lidocaine + bupivacaine + clonidine: Submucosal injection of 1.5 mL into each tonsillar fossa prior to performing tonsillectomy with one of three injections.
  C - lidocaine (1%) + bupivacaine (0.5%) + clonidine (25mcg)
Period: Overall Study
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Started | 40 | 40 | 40
Completed | 34 | 37 | 36
Not Completed | 6 | 3 | 4
Not completed — Injection performed after tonsillectomy | 2 | 0 | 1
Not completed — Incomplete Data | 4 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Median (Full Range); unit: years] | 6 [5 to 9] | 7 [5 to 11] | 8 [5 to 12] | 7 [5 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 23 | 67
  Male | 16 | 20 | 17 | 53
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Post-operative Doses of Analgesics.
Description: The total number of intravenous fentanyl doses given PACU which will be compared between the three randomized groups (arms)
Time Frame: Post-operative thru day 7
Population: Number of patients randomized to each group
Measure: Median (Full Range); unit: number of doses
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
number of doses | 12 [9 to 15] | 12 [10 to 16.5] | 14 [9 to 16.8]

2. Secondary Outcome: Median Number of Pain Medication Doses
Description: The median number of intravenous fentanyl doses administered in the PACU due to pain
Time Frame: in recovery room
Population: per group doses
Measure: Median (Full Range); unit: number of doses
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
number of doses | 3.0 [3.0 to 5.0] | 3 [2 to 4] | 3 [2 to 4]

3. Secondary Outcome: Total Time Until Discharge From Hospital.
Time Frame: Day of Surgery
Measure: Median (Full Range); unit: minutes
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
minutes | 122 [90 to 188] | 111 [81 to 142] | 120 [79 to 175]

4. Secondary Outcome: Mean Visual Analog Scale Pain Number.
Description: Visual analog pain scale range is 0-10 with 0=no pain and 10 = worst pain ever
Time Frame: in recovery room; post-operative days 1,3,5 & 7
Measure: Mean (Full Range); unit: pain score
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
pain score
  In recovery room | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]
  day 1 | 3 [2 to 6] | 4 [3 to 5] | 5 [4 to 5.2]
  day 3 | 3 [1 to 3.5] | 2.5 [2 to 4] | 3 [2 to 5]
  day 5 | 3 [1.5 to 5] | 2 [1 to 5] | 3 [2 to 6]
  day 7 | 2.5 [1 to 3.2] | 2 [1 to 5] | 2 [1 to 4]

5. Secondary Outcome: Number and Percent of Participants Able to Tolerate Only Liquids
Description: The number and percent of patients whose post-operative diet has advanced to liquids only on post-op days 1, 3, 5 & 7
Time Frame: post-operative days 1,3,5 & 7.
Population: per group data
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
Participants
  post-op day 1 | 16 | 33 | 30
  post-op day 3 | 8 | 13 | 23
  post op day 5 | 13 | 10 | 19
  post op day 7 | 6 | 11 | 10

6. Secondary Outcome: Number and Percent of Participants Able to Tolerate Only a Soft Diet
Description: The number and percent of patients whose post-operative diet has only advanced to a soft diet on post-operative days 1, 3, 5 & 7
Time Frame: post-operative days 1,3,5 & 7.
Population: per group diet
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
Participants
  post-op day 1 | 26 | 22 | 26
  post-op day 3 | 18 | 26 | 18
  post op day 5 | 13 | 17 | 18
  post op day 7 | 13 | 10 | 14

7. Secondary Outcome: Number and Percent of Participants Able to Tolerate a Regular Diet
Description: The number and percent of patients whose post-operative diet has to a regular diet on post-operative days 1, 3, 5 & 7
Time Frame: post-operative days 1,3,5 & 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
Number analyzed (Participants) | 40 | 40 | 40
Participants
  post-op day 1 | 7 | 4 | 1
  post-op day 3 | 18 | 8 | 12
  post op day 5 | 21 | 18 | 14
  post op day 7 | 24 | 26 | 22

ADVERSE EVENTS:
Time Frame: Each patient was followed for adverse events for the duration they were in the study and up to their post-operative visit at 3 weeks post-surgery.
Description: We used the same definition.
Arm/Group | Normal Saline | Lidocaine (1%) + Bupivacaine 0.5% | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 4/40 | 6/40 | 6/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=40) | Lidocaine (1%) + Bupivacaine 0.5% (N=40) | Lidocaine 1% + Bupivacaine o.5% + Clondine 25mcg (N=40)
Dehydration (General disorders) | 1 (1) | 3 (3) | 3 (3)
Emergency Department admission (General disorders) | 0 (0) | 1 (1) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1)
Lingual nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Severe pain (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No